CLINICAL TRIAL: NCT04704596
Title: Lung Ultrasound Versus Dynamic Lung Compliance to Detect the Optimum PEEP After Alveolar Recruitment for Patients Undergoing Laparoscopic Gastric Sleeve Surgery, Randomized Clinical Trial
Brief Title: Lung Ultrasound Versus Dynamic Lung Compliance to Detect the Optimum PEEP After Alveolar Recruitment for Patients Undergoing Laparoscopic Gastric Sleeve Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amin Mohammed Alansary Amin Ahmed Helwa, Assistant professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FMASU R 127/2020
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Mechanical Ventilation During Anesthesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dynamic lung compliance for detection of optimum PEEP (Active Comparator): detection of optimum PEEP by measurement of the dynamic lung compliance (by the ventilator machine) after lung recruitment
  Interventions: Device: anesthesia ventilator machine
- Lung ultrasound for detection of the optimum PEEP (Active Comparator): Lung ultrasound will be used to detect the optimum PEEP after lung recruitment
  Interventions: Device: lung ultrasound

INTERVENTIONS:
Device: anesthesia ventilator machine — dynamic lung compliance measurements will be used for detection of the optimum PEEP after alveolar recruitment
  Arms: dynamic lung compliance for detection of optimum PEEP
Device: lung ultrasound — lung ultrasound views will be used for detection of the optimum PEEP after alveolar recruitment
  Arms: Lung ultrasound for detection of the optimum PEEP

SUMMARY:
The aim of this study is to evaluate The role of transthoracic lung US as a clinical tool in Comparison to dynamic lung compliance for detection of optimum PEEP for obese patients undergoing laparoscopic gastric sleeve surgery.

ELIGIBILITY:
Inclusion Criteria:

* physical status American Society of Anesthesiologist(ASA) I or II

Exclusion Criteria:

* Patients refuse ASA physical status more > II
* Patients with pre-existing significant pulmonary disease with abnormalities in spirometry, previous lung surgery, home oxygen therapy and signiﬁcant cardiac dysfunction.
* Patients with pulmonary hypertension.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
detection of the optimum PEEP which is measured in mmHg | intraoperative period
  the optimum PEEP will be detected after alveolar recruitment either by dynamic lung compliance or by lung ultarsound views

SECONDARY OUTCOMES:
prevention of postoperative pulmonary complications | 1st 24 hour
  patients will be monitored for detection of postoperative pulmonary complictaios as atelectasis , pneumothorax , respiratory failure

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes